CLINICAL TRIAL: NCT00420914
Title: Strategies for Transfusion of Platelets (SToP) [Formerly Titled "Evaluation of the Hemostatic Efficacy and Platelet Utilization Rates of Low Versus Standard Dose Platelet Therapy"]
Brief Title: Strategies for Transfusion of Platelets (SToP)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped at the request of the Data Safety Monitoring Board for safety reasons.
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); Haukeland University Hospital (Other); Ottawa Hospital Research Institute (Other); Cedars-Sinai Medical Center (Other); University Health Network, Toronto (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SToP Study
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Platelets; Dose; Bleeding
MeSH Terms: conditions — Thrombocytopenia; Hemorrhage | interventions — Blood Transfusion

INTERVENTIONS:
Procedure: low dose of 2.25 x 10^11 platelets/transfusion (range 1.5 to 2.9)

SUMMARY:
To evaluate the hemostatic efficacy of a low dose platelet transfusion strategy compared to a standard dose platelet transfusion strategy.

DETAILED DESCRIPTION:
BACKGROUND:Platelet transfusions play a major role in the management of thrombocytopenic patients. Platelet transfusions may be given either in the absence of hemorrhage (prophylactic transfusions), or to control bleeding (therapeutic transfusions). Prophylactic platelet transfusion therapy is most commonly used in patients with decreased marrow platelet production (hypoproliferative thrombocytopenia) and accounts for the majority of platelets transfused to these patients. As platelet use continues to increase at a rate disproportionately higher than that of red cells, it is important to identify the most cost-effective strategies for providing platelet support. The two most important factors - within the control of the ordering physician - that will significantly influence the total amount of platelets transfused are:

1. the prophylactic platelet transfusion "trigger" selected for transfusion;
2. the number of platelets given per transfusion. The optimal quantity of platelets to be used per transfusion remains a highly controversial subject. No prospective platelet transfusion trials have been performed in which patients are randomized to an assigned platelet dose throughout their period of thrombocytopenia to evaluate the effects of different doses on transfusion outcomes.

INTRODUCTION: A randomized prospective platelet dose trial is proposed to determine a safe, efficient, and cost-effective dosing strategy for transfusing platelets. The trial is designed to answer two fundamental questions: 1) Are low dose platelet transfusions not inferior to standard dose platelet transfusion for patients with chemotherapy induced thrombocytopenia as measured by the frequency of WHO bleeding Grade 2 or greater; and 2) How does the dose of platelets transfused affect the interval between platelet transfusion events, and, thereby, the total number of platelets transfused?

GENERAL OBJECTIVE: To evaluate the hemostatic efficacy of low dose platelet transfusions.

PRIMARY OBJECTIVE: This will be a non-inferiority study designed to determine if low dose prophylactic platelet transfusions can be transfused to patients with chemotherapy induced thrombocytopenia without an increase in the frequency of WHO bleeding (Grade 2 or greater ) when compared to the current transfusion strategy of using standard dose platelet products.

The low dose platelet transfusions will be targeted at 2.25 x 10^11 platelets/transfusion (range 1.5-2.9 x 10^11/product).

The standard dose platelet transfusions will be targeted at 4.5 x 10^11 platelets/transfusion (range 3.0-6.0 x 10^11/ product)

STUDY DESIGN: This will be a multicenter prospective randomized controlled trial in which eligible patients will be randomized to receive low dose or standard dose prophylactic platelet transfusions. Patients will be transfused prophylactically using a transfusion trigger of a platelet count equal to or below a level of 10 x 10^9/L (10,000/uL)or at a higher trigger (dependant on transfusion guidelines set by individual institutions).

Clinical evidence of bleeding will be assessed daily according to the WHO classification of bleeding. Study personnel involved in the daily hemostatic assessments of patients will be blinded as to the patient's randomization assignment. The grade of bleeding will be assigned using an Adjudication Committee blinded to the treatment that each patient is receiving. Each patient will be followed throughout their period of thrombocytopenia.

A Data and Safety Monitoring Board (DSMB) has been established and is comprised of two hematologists not associated with the study, one critical care physician, and a biostatistician. Three of these individuals have experience serving on Data Safety Monitoring Boards and all have expertise in clinical research methodology. The DSMB will receive and review any adverse events and regular reports. The information on the report will be blinded by designating treatment groups as A or B.

STRATIFICATION: There will be two levels of stratification in this study. The first level of stratification will be by center as there will be center differences in the chemotherapy and bone marrow or stem cell transplant protocols used. The second level of stratification will be by diagnostic grouping: bone marrow/stem cell transplant; and non transplant patients.

TREATMENT ALLOCATION: Eligible patients who have given written consent, will be randomized to a treatment arm when they require their first prophylactic platelet transfusion.

INTERVENTION: Patients will be randomized to one of two prophylactic platelet transfusion strategies either low dose or standard dose.

At the time of each platelet transfusion, a platelet count will be performed on the product and the weight of the platelet bag will be recorded so that the absolute number of platelets given with each platelet transfusion can be calculated. Either apheresis platelets or whole blood derived platelet concentrates will be used to achieve the required platelet dose based on product availability or the preferences of the patient's physician.

PERIOD OF FOLLOW-UP: Study patients will be followed throughout their period of thrombocytopenia until bone marrow recovery has occurred (with a platelet count of ≥ 50 x10^9/L (50,000/uL) or the patient has been on the study for 30 days, withdraws consent, dies or is discharged from hospital or to a setting that does not allow for daily assessment of bleeding.

SERIOUS ADVERSE EVENTS: WHO Grade 3 or 4 bleeding will be considered a serious adverse event and will be monitored throughout the study. These serious adverse events will be reported to the data coordinating center and to the relevant IRB within 24 hours.

ANALYSIS OF PRIMARY OBJECTIVE: There will be two analyses performed: the first will compare the proportion of patients in each treatment group that have Grade 2 or greater bleeding: the second will be a recurrent event analysis which uses a strategy that includes the proportion of patients who bleed, the numbers of bleeds that occur and the timing of the bleed (i.e. whether it occurs early or late during the period of thrombocytopenia).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypoproliferative thrombocytopenia who are expected to have a platelet count of ≤ 10,000/µL (10x10^9/L) for ≥ 10 days (Note: the prophylactic platelet trigger may be higher than10,000/µL (10x10^9/L) in some participating institutions; however, the patient will still be eligible for participation as long as they are expected to be thrombocytopenic for 10 days)
* Must be an inpatient.
* Weight between 40 and 100 kg.

Exclusion Criteria:

* Diagnosis of promyelocytic leukemia.
* A history or current diagnosis of immune thrombocytopenia (ITP), thrombotic thrombocytopenia (TTP), or hemolytic uremia syndrome (HUS).
* Evidence of ≥ WHO Grade 2 bleeding while being assessed for the study entry.
* Patients who will receive bedside Leukoreduced platelet transfusions.
* Patients who are pregnant.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Daily hemostatic assessments will be conducted to determine presence of WHO Grade 2 bleeding or greater.

SECONDARY OUTCOMES:
Number of platelets transfused during a defined period of thrombocytopenia
Number of platelet transfusion events(frequency)
Number of platelets transfused and frequency per thrombocytopenic day
Mean duration of thrombocytopenia
Percentage of days at risk of bleeding
Differences in the severity of bleeding between treatment groups
Correlation between the actual platelet dose given per transfusion for each patient and bleeding on the day following transfusion
Correlation between the actual number between the actual number of platelets transfused/kg body weight for each patient and bleeding on the day following transfusion
Pre- and post-transfusion bleeding grade in response to the dose of therapeutic platelets transfused
Surrogate outcomes for hemostatic efficacy including death due to bleeding as the primary and contributory cause of mortality
Platelet transfusion given above trigger
Platelet transfusion more often than once a day
Platelet transfusion given above their assigned dose in each case because of >/= WHO Grade 2 bleeding
Number of platelets transfused
Frequency of transfusions and duration of transfusions given because of bleeding
Total number of RBC transfusions
The mean per thrombocytopenic day for each patient
Platelet response (pre-transfusion platelet counts, post-transfusion platelet counts, platelet increments, and corrected platelet count increments (at 1 and/or 24 hours)
Cost analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Heddle, MSc., FCSMLS(D), Principal Investigator — McMaster University
Locations (6):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Heddle NM, Cook RJ, Tinmouth A, Kouroukis CT, Hervig T, Klapper E, Brandwein JM, Szczepiorkowski ZM, AuBuchon JP, Barty RL, Lee KA; SToP Study Investigators of the BEST Collaborative. A randomized controlled trial comparing standard- and low-dose strategies for transfusion of platelets (SToP) to patients with thrombocytopenia. Blood. 2009 Feb 12;113(7):1564-73. doi: 10.1182/blood-2008-09-178236. Epub 2008 Dec 24. PMID 19109560